CLINICAL TRIAL: NCT04866030
Title: Drug Utilization Study With Intuniv® in Australia
Brief Title: Drug Use Study With Intuniv® in Australia
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP503-803; EUPAS40684 (Registry Identifier: EU PAS Registry)
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NostraData Database: All prescriptions for Intuniv available in the NostraData database in Austrialia will be analyzed in this study.
- Physician Survey: Physician will collect medical record data of 100 participants who have been prescribed Intuniv at least once during the study period to treat participants with ADHD.

SUMMARY:
This study will evaluate and analyze prescribing behaviors of physicians and determine whether Intuniv was correctly prescribed in Australia.

DETAILED DESCRIPTION:
This is a drug utilization study using retrospective database analysis where study will combine data from two sources of patient-level drug utilization data for Intuniv:

i) NostraData database: longitudinal participant level prescription database ii) Physician survey: de-identified participant data provided by representative physicians in Australia

In the NostraData database, actual prescription data are collected, which allows generation of information on drug usage. However, these prescription data do not contain patient variables such as age and indication needed to monitor potential off-label use. Therefore, these data must be supplemented with another data source. The physician survey will provide the data not included in the NostraData database.

ELIGIBILITY:
Inclusion Criteria:

* Is indicated for the treatment of ADHD in children and adolescents 6 to 17 years old, as monotherapy.
* Must be used as a part of a comprehensive ADHD treatment programme, typically including psychological, educational and social measures.

Exclusion Criteria:

* Use for participants with a diagnosis other than ADHD.
* Use for children less than 6 years of age.
* Use in adults (greater than or equal to [>=] 18 years of age)
* Prescribed overdose greater than (>) 7 milligram per day (mg/day) for participants > 12 years, or > 4 mg/ day for children lesser than or equal to (<=) 12 years.
* If monotherapy with Intuniv, no prior treatment with stimulants or atomoxetine.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants who have been prescribed Intuniv at least once during the reporting period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants Based on Indication of Use of Intuniv | Up to 3 years
  Number of Participants Based on Indication of Use of Intuniv will be assessed.
Number of Participants with Presence/Absence of Contraindications | Up to 3 years
  Number of participants with presence/absence of contraindications will be assessed.

SECONDARY OUTCOMES:
Number of Participants Based on Patterns of Drug Use | Up to 3 years
  Patterns of drug use will include daily dose, first time user, repeat user, treatment duration, treatment gaps, discontinuation of ADHD therapy and switch of therapy, co-prescriptions of ADHD medication.
Number of Participants Stratified by Prescriber Information Based on Physician Survey | Up to 3 years
  Participants will be stratified based on prescriber information which include specialty, graduation year, gender, location, and region.
Frequency of Weight Monitoring of Participants by Physician | Up to 3 years
  Frequency of weight monitoring of participants by physician will be reported.
Frequency of Blood Pressure Monitoring of Participants by Physician | Up to 3 years
  Frequency of blood pressure monitoring of participants by physician will be reported.
Frequency of Heart Rate Monitoring of Participants by Physician | Up to 3 years
  Frequency of heart rate monitoring of participants by physician will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Site, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/609017abf89629001e47b500